CLINICAL TRIAL: NCT07396831
Title: Safety of Retina Surgery Without Postoperative Eye Drops
Brief Title: Necessity of Post-operative Eye Drops
Status: Terminated | Type: Observational
Why Stopped: PI left institution. No new PI.
Sponsor: Loma Linda University (Other)
Responsible Party: Sponsor
Other Study IDs: 5230480
Record Dates: First submitted 2026-02-02; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Pars Plana Vitrectomy; Scleral Buckling; Surgical Outcomes; Infection Prophylaxis
Keywords: Pars plana vitrectomy; Scleral buckling; Infection prophylaxis; Topical antibiotics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this clinical study is to determine if antibiotic eye drops are needed after retinal surgery to prevent infection. Currently, patients are prescribed antibiotic eye drops to use for several weeks after they undergo retina surgery. The main question that we are trying to answer is:

- Are postoperative eye drops necessary to prevent eye infections after retina surgery? Patients will still receive steroid drops after their surgery to control inflammation. Additionally, patients will have regular follow up with their eye surgeon to monitor for the signs and symptoms of eye infection.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing Pars plana vitrectomy and/or scleral buckling

Exclusion Criteria:

* Patients younger than 18
* Patients undergoing Pars plana vitrectomy for endophthalmitis
* Patients having combined intraocular lens and vitrectomy surgery
* Patients that received a cornea scrape during surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients from a single vitreoretinal surgeon at Loma Linda University Medical Center.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2024-04-09 (Actual); Primary Completion 2025-12-22 (Actual); Study Completion 2025-12-22 (Actual)

PRIMARY OUTCOMES:
Presence of endophthalmitis | 30 days
  The primary outcome of this study is the presence of endophthalmitis 30 days after pars plana vitrectomy and/or scleral buckling without the use of post-operative antibiotics.

CONTACTS AND LOCATIONS:
Overall Officials: Bailey Shen, Doctor of Medicine, Principal Investigator — Loma Linda University Eye Institute
Locations (1):
- Loma Linda University Eye Institute, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Only IPD used in the results publication will be shared

REFERENCES:
- [Background] Dave VP, Pathengay A, Schwartz SG, Flynn HW Jr. Endophthalmitis following pars plana vitrectomy: a literature review of incidence, causative organisms, and treatment outcomes. Clin Ophthalmol. 2014 Oct 31;8:2183-8. doi: 10.2147/OPTH.S71293. eCollection 2014. PMID 25382968